CLINICAL TRIAL: NCT03221660
Title: Clinical Investigation of the F-Composite 2 System in Direct Filling Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 621211
Record Dates: First submitted 2017-07-13; First posted 2017-07-18 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries; Unsatisfactory or Defective Restoration of Tooth
Keywords: filling material, polymerization
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- F-Composite 2 system (Experimental): Tooth (teeth) affected by dental caries or with an existing defective filling will be restored using the F-Composite 2 system.
  Interventions: Device: F-Composite 2 system

INTERVENTIONS:
Device: F-Composite 2 system — Procedures will be done using local anesthesia (if the patients wants that). The cavity is prepared according to the principles of the adhesive technique. First the adhesive will be applied and polymerized, afterwards the flowable resin-based restorative material will be applied and polymerized and then the sculptable resin-based restorative material will be applied and polymerized; all materials will be light-cured within short time with an experimental curing light.

SUMMARY:
The objective of this study is to evaluate the clinical performance of F-Composite 2 system in Class I and Class II cavities in permanent teeth.

The materials of the system can be polymerized in short time with a curing light which is part of the system.

The study will be carried out as a prospective study, with evaluation of the restorations after 7-10 days (baseline), at 6 months, at 12 months, at 24 months and 60 months according to defined criteria.

ELIGIBILITY:
Inclusion Criteria:

* Indication for direct filling of Class I or II with permanent premolars or permanent molars
* replacement of insufficient fillings (e.g., due to edge caries, filling fracture, Lack of quality of the surface, lack of aesthetics, undesirable filling material, leaky edge, edge gap, etc.)
* extensive primary caries
* Vital tooth (cold test)
* One-, two- or three-surface fillings in the lateral tooth area, with a maximum of 25% single-faced (Class I) with antagonists.
* The occlusal area of the filling must be at least 1/3 of the total area of the filling tooth. This criterion is estimated.
* Patient wishes to receive care within the framework of the study (written consent after detailed elucidation and study of patient information).
* Maximum of 2 restorations per patient.
* Preoperative complaints on the tooth to be restored (maximum 3 on visual Analog scale (0 = complaint-free, 10 = maximum possible pain) to temperature or bite sensitivity
* Sufficient language skills

Exclusion Criteria:

* Unfinished hygiene phase or poor oral hygiene
* Sufficient draining of the operating field is not possible
* Patients with proven allergy to one of the ingredients of the materials used
* Patient has allergies to local anesthetic agents Ultracain DS (active substance: articaine; Vasoconstrictor), if anesthesia is desired
* Patients with severe systemic diseases
* Devital or pulpitic teeth
* Periodontal insufficiency
* Supplements with cusp attachments
* open side bite
* missing antagonist
* Indication for direct capping
* Pregnancy (women of childbearing age receive a free pregnancy test for self application, the negative result of which is shown with her confirmed consent).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Enggist, Dr, Principal Investigator — dentist internal clinic
Locations (1):
- Ivoclar Vivadent, Schaan, Liechtenstein

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: teeth
Groups:
- F-Composite 2 System: 75 teeth affected by dental caries or with an existing defective filling were restored using the F-Composite 2 system. 25 participants received two fillings and 25 received only one filling.
  F-Composite 2 system: Procedures was done using local anesthesia (if the patients wants that). The cavity was prepared according to the principles of the adhesive technique. First the adhesive was applied and polymerized, afterwards the flowable resin-based restorative material was applied and polymerized. Then the sculptable resin-based restorative material was applied and polymerized. All materials were light-cured within short time with an experimental curing light.
Period: Overall Study
Arm/Group | F-Composite 2 System
Started | 50; 75 teeth
Completed | 42; 60 teeth
Not Completed | 8; 15 teeth

BASELINE CHARACTERISTICS:
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 50
Number analyzed (Teeth) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: Teeth]
  Liechtenstein | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Restored Teeth With Postoperative Sensitivity
Description: The postoperative sensitivity is assessed by tests with thermal stimuli and occlusal forces (during biting) determined by VAS (Visual Analog Scale, from 0 "no pain" to 10 "maximum pain") following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable".
  A maximum of 10% postoperative hypersensitivities are defined as acceptable after one month.
Time Frame: 1 month
Measure: Number; unit: percentage restored hypersensitive teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 50
Number analyzed (Teeth) | 75
percentage restored hypersensitive teeth | 7

2. Secondary Outcome: Number of Restored Teeth With Loss of Vitality
Description: The loss of vitality of restored teeth is assessed by a cold stimuli test (cotton pellet and refrigerating spray) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable".
  A maximum of 1 tooth with loss of vitality within 12 months is determined to be acceptable.
Time Frame: 12 months
Population: The participants analyzed and number of teeth (units) analyzed differs from the number of participants and units assigned to the arm as 1 participant with 2 fillings did not attend the 12-month recall.
Measure: Number; unit: teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 49
Number analyzed (Teeth) | 73
teeth | 0

3. Secondary Outcome: Replacement of Filling
Description: maximum of 3 fillings which have to be replaced due to a lack of quality after 2 years
Time Frame: 2 years
Measure: Number; unit: replaced fillings due to quality
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 49
Number analyzed (Teeth) | 73
replaced fillings due to quality | 0

4. Other Pre Specified Outcome: FDI 1 Surface Luster, FDI Score 1-5
Description: assessed on patient teeth (comparing surface of filling with enamel) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 60 months
Population: 7 patients with 12 restorations were not able to attend final recall after 5 years. 3 restorations were replaced because patient suffered from hypersensitivoity on bitting/chewing. 60 from the initial 75 restoratons were analyzed
Measure: Number; unit: Teeth
Units Other Than Participants: teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 42
Number analyzed (teeth) | 60
Teeth
  FDI 1 Surface Luster, FDI Score 1 | 6
  FDI 1 Surface Luster, FDI Score 2 | 45
  FDI 1 Surface Luster, FDI Score 3 | 9
  FDI 1 Surface Luster, FDI Score 4-5 | 0

5. Other Pre Specified Outcome: FDI 2 Surface Staining, FDI Score 1-5
Description: assessed on patient teeth by checking surface staining of restoration following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 60 month
Population: as for outcome 4
Measure: Number; unit: teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 42
Number analyzed (Teeth) | 60
teeth
  FDI 2 Surface Staining, FDI Score 1 | 42
  FDI 2 Surface Staining, FDI Score 2 | 17
  FDI 2 Surface Staining, FDI Score 3 | 1
  FDI 2 Surface Staining, FDI Score 4-5 | 0

6. Other Pre Specified Outcome: FDI 3 Translucency, FDI Score 1-5
Description: assessed on patient teeth by checking differences in shade and translucency following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 60 month
Population: as for outcome 4
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 42
Number analyzed (Teeth) | 60
Teeth
  FDI 3 Translucency, FDI Score 1 | 43
  FDI 3 Translucency, FDI Score 2 | 17
  FDI 3 Translucency, FDI Score 3-5 | 0

7. Other Pre Specified Outcome: FDI 5 Retention/Fracture of Restorations, FDI Score 1-5
Description: assessed on patient teeth (checking irestorations for fractures, cracks, small hairline cracks, chip fractures, material damage) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 60 month
Population: as for outcome 4
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 42
Number analyzed (Teeth) | 60
Teeth
  FDI 5 Fracture of material and retention, FDI Score 1 | 51
  FDI 5 Fracture of material and retention, FDI Score 2 | 4
  FDI 5 Fracture of material and retention, FDI Score 3 | 5
  FDI 5 Fracture of material and retention, FDI Score 4-5 | 0

8. Other Pre Specified Outcome: FDI 6 Marginal Adaption, FDI Score 1-5
Description: assessed on patient teeth (checking for hamonious outline, gaps and white/discolored lines)) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 60 month
Population: as for outcome 4
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 42
Number analyzed (Teeth) | 60
Teeth
  FDI 6 Marginal Gap, FDI Score 1 | 49
  FDI 6 Marginal Gap, FDI Score 2 | 9
  FDI 6 Marginal Gap, FDI Score 3 | 2
  FDI 6 Marginal Gap, FDI Score 4-5 | 0

9. Other Pre Specified Outcome: FDI 10 Patient's View, FDI Scire 1-5
Description: assessed by discussion with the patient (satisfied with esthetics and function) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 60 month
Population: as for outcome 4
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 42
Number analyzed (Teeth) | 60
Teeth
  FDI 10 Patient's View, FDI Score 1 | 60
  FDI 10 Patient's View, FDI Score 2-5 | 0

10. Other Pre Specified Outcome: FDI 11 Postoperative Hypersensitivity and Tooth Vitality, FDI Scores 1-5
Description: Hypersensitivity was assessed by tests with thermal stimuli and occlusal forces (during biting) determined by VAS (Visual Analog Scale) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable".
  Tooth vtality assessed by a cold stimuli test on the patient teeth (cotton pellet and refrigerating spray) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 60 month
Population: as for outcome 4
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 42
Number analyzed (Teeth) | 60
Teeth
  FDI 11 Postoperative hypersensitivity and tooth vitality, FDI Score 1 | 60
  FDI 11 Postoperative hypersensitivity and tooth vitality, FDI Score 2-5 | 0

11. Other Pre Specified Outcome: FDI 12 Recurrence of Caries (CAR), Erosion, Abfraction, FDI Scores 1-5
Description: assessed on patient teeth (primary caries, areas of demineralization erosion or abfraction)) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 60 month
Population: as for outcome 4
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 42
Number analyzed (Teeth) | 60
Teeth
  FDI 12 Recurrence of Caries (CAR), erosion, abfraction, FDI Score 1 | 59
  FDI 12 Recurrence of Caries (CAR), erosion, abfraction, FDI Score 2 | 1
  FDI 12 Recurrence of Caries (CAR), erosion, abfraction, FDI Score 3-5 | 0

12. Other Pre Specified Outcome: FDI 13 Tooth Integrity, FDI Scores 1-5
Description: assessed on patient teeth by checking tooth integrity (looking for enamel cracks, tooth fractures) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 60 month
Population: as for outcome 4
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | F-Composite 2 System
Number analyzed (Participants) | 42
Number analyzed (Teeth) | 60
Teeth
  FDI 13 Tooth integrity, FDI Score 1 | 58
  FDI 13 Tooth integrity, FDI Score 2-3 | 0
  FDI 13 Tooth integrity, FDI Score 4 | 1
  FDI 13 Tooth integrity, FDI Score 5 | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | F-Composite 2 System
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 4/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-Composite 2 System (N=50)
Long-term hypersensitivity (General disorders) | 3 (3) — Fillings needed to be replaced due to long-term hypersensitivity. It is generally related to this type of clinical procedure and might also be dependent on the applied light intensity, the used adhesive or the backstory of the tooth.
Unrelated: Fracture of disto-lingual cusp next to study tooth (General disorders) | 1 (1) — The fracture was partly at the border to the study restoration. But the restoration remained intact and was available for the 60-month recall. This adverse event is unrelated to the clinical procedure and to the investigational device itself.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT03221660/Prot_SAP_000.pdf